CLINICAL TRIAL: NCT06928727
Title: Ocular Characteristics in Patients With Craniosynostosis
Acronym: COPACA
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2025_843_0075
Record Dates: First submitted 2025-04-08; First posted 2025-04-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Craniosynostosis; Strabismus; Intracranial Hypertension; Amblyopia
Keywords: Craniosynostosis; strabismus; amblyopia; intracranial hypertension
MeSH Terms: conditions — Craniosynostoses; Strabismus; Intracranial Hypertension; Amblyopia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Craniosynostosis are cranial deformations due to the premature closure of one or more cranial sutures. These deformations affect approximately one in 2.500 births. In most cases, craniosynostoses are isolated with unknown (non syndrome). On the other hand, 20% of these deformations are associated with other concentration (syndrome).

Craniosynostosis has morphological (associated dysmorphism) and functional (growth conflict between the skull and the brain) repercussions. Ophthalmological disorders are frequent: refractive disorders, oculomotor disorders, optic nerve damage, sensory damage.

This retrospective study aims to describe the ocular clinical characteristics associated with craniosynostosis in patients followed at the Amiens University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of craniostenosis

Exclusion Criteria:

* Posterior plagiocephalia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with craniosynostosis followed at the Amiens University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Rate of strabismus and amblyopia | 6 months
  Rate of strabismus and amblyopia

SECONDARY OUTCOMES:
Rate of intracranial hypertension | 6 months
  Rate of intracranial hypertension

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No